CLINICAL TRIAL: NCT01644981
Title: Prospective Study on Plasma Pro-endothelin-1 in Predicting Bronchopulmonary Dysplasia
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 1.3 07.10.2011
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VLBW infants
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling

SUMMARY:
Serial quantitative measurements of plasma pro-endothelin-1 concentrations in very preterm infants. Comparing pro-endothelin-1 with established clinical indices of bronchopulmonary dysplasia (BPD). Hypothesis: Pulmonary-vascular remodeling in infants developing BPD is directly related to circulating pro-endothelin-1, which therefore serves as surrogate marker of BPD.

ELIGIBILITY:
Inclusion criteria:

* Very preterm infants born before 32 weeks gestational age

Exclusion criteria:

* Severe fetal malformation, congenital heart defect, inborn syndrome, cardiomyopathy, fetal hydrops

Ages: 2 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants born before 32 weeks gestational age
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
duration of supplemental oxygen requirement | 36 weeks postmenstrual age
  Bronchopulmonary dysplasia

SECONDARY OUTCOMES:
duration of respiratory pressure support | during hospitalisation
  respiratory pressure support either mechanical and/or nCPAP (days)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Wellmann, MD, Principal Investigator — University Hospital Zurich, Division of Neonatology
Locations (1):
- University Hospital Zurich, Division of Neonatology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided